CLINICAL TRIAL: NCT02381808
Title: Study on Potential Biomarkers Associated With Clinical Phenotype of EGFR-TKIs in No-small Cell Lung Cancer in China
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Guangdong Association of Clinical Trials (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: CTONG1502; BI1200.250 (Other Grant/Funding Number: Boehringer Ingelheim)
Record Dates: First submitted 2015-03-05; First posted 2015-03-06 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Frozen tissue or tissue block
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To understand 295 gene mutation mutation status (include EGFR, HER2, KRAS, BRAF, PIK3CA,ect) by deep sequencing in Chinese patients with pulmonary adenocarcinoma and their relationships with the patients' clinical features (including sex, age, smoking history and adenocarcinoma subtype), specify the predictive significance of the genes mutations for new targeted therapies in NSCLC patients, and better understand the molecular mechanism drug resistance to EGFR-TKIs.

DETAILED DESCRIPTION:
This study is prospective to identify biomarkers to resistant to afatinib，gefitinib and erlotinib in non-small cell lung cancer patients. Mutations of whole exon of 295 gene are analysed by deep sequencing in Chinese patients with non-small cell lung cancer and their relationships with the patients' clinical features (including sex, age, smoking history and adenocarcinoma subtype), specify the predictive significance of the genes mutations for new targeted therapies in NSCLC patients, and better understand the molecular mechanism drug resistance to EGFR-TKIs.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years,both male and female
* Histologically confirmed patients with pulmonary adenocarcinoma (Stage I-IV)
* ECOG 0-2
* Patients with enough paraffin tissue specimens or fresh tissue for detection
* Quality of the DNA extracted from the tissue samples ensures that the DNA can be used in DNA sequencing
* Subjects who provide detailed clinical and follow-up information

Exclusion Criteria:

* Patients with other tumors
* Patients suffering from other serious diseases like infectious diseases (viral hepatitis, HIV,etc)
* Pregnant women shall be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NSCLC (SageI-IV)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-06-24 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Potential predictive biomarker to resistant to afatinib | baseline
  Mutations of whole exon of 295 gene are analysed by deep sequencing in Chinese patients with NSCLC and their relationships with the patients' clinical features , specify the predictive significance of the genes mutations for new targeted therapies in NSCLC patients, and better understand the molecular mechanism drug resistance to EGFR-TKIs

CONTACTS AND LOCATIONS:
Overall Officials: China China, Study Chair — Guang general hospital,Guangzhou, Guangdong, China, 510080
Locations (1):
- Guangdong General Hospital & Guangdong Academy of Medical Sciences, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided